CLINICAL TRIAL: NCT04341415
Title: Randomized Double Blinded Monocentric Clinical Trial to Assess the Impact of Auricular Vagus Nerve Neuromodulation in COVID-19 Positive Inpatients Outcome.
Brief Title: Impact of Auricular Vagus Nerve Neuromodulation on COVID-19 Positive Inpatients Outcome
Acronym: SOS-COVID19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion stopped at 50% after interim analysis: primary efficacy endpoint not significant
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRN_2020_8
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: Non-invasive Neuromodulation; Vagus Nerve
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants and the care providers will not know the arm of randomization. Only the principal investigator who will perform the intervention will know the type of intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular neuromodulation (Experimental)
  Interventions: Procedure: Auricular neuromodulation
- Control (Sham Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Auricular neuromodulation — The pose is carried out by the principal investigator, alone, without the presence of the nursing staff in the room.
  Ear disinfection and sterile neuromodulation needle placement (service protocol with Chlorhexidine) Placement of 4 semi-permanent Classic needles (SEDATELEC®) on each ear flap at the level of the concha (innervated by the vagus nerve) according to an order and a precise location (4 cardinal points conch), i.e. 8 needles per patient.
  Compress soaked with Oxygenated water on the concha (to stop potential bleeding).
  Placing an opaque dressing on the ear and a non-occlusive Band-Aid
  Other Names: VERUM
  Arms: Auricular neuromodulation
Procedure: Control — The pose is carried out by the principal investigator, alone, without the presence of the nursing staff in the room.
  Ear disinfection and sterile manipulation without needle placement (service protocol with Chlorhexidine) No needle laying but only sterile disinfection and pressure over the 4 putative locations with the sterile plastic tip (without the needle).
  Compress soaked with Oxygenated water on the concha. Placing an opaque dressing on the ear and a non-occlusive Band-Aid.
  Other Names: SHAM
  Arms: Control

SUMMARY:
The COVID-19 pandemic has already overwhelmed the sanitary capacity. Additional therapeutic arsenals, albeit untested in the given context but previously proven to be efficacious in a related clinical context, that could reduce the morbidity rate are urgently needed.

A decrease of Heart Rate Variability (HRV) is a validated bad prognosis marker in sepsis and acute respiratory distress syndrome.

In contrast, auricular vagus nerve stimulation was proven not only to increase HRV values in healthy Humans, but also to reduce sepsis and increase survival, both significantly, in experimental models.

Moreover, the heavy viral infection within the brainstem of deceased patients suggests that the neuroinvasive potential of SARS-CoV2 is likely to be partially responsible for COVID-19 acute respiratory failure and may bear relevance in tailoring future treatment modalities.

Interestingly, the vagus nerve (or tenth cranial nerve) connects bidirectionally the brainstem to various internal organs including the lung and to one external organ, namely, the outer ear.

Hence, the impact of auricular vagus nerve stimulation through semi-permanent needles will be studied, mostly used so far for pain alleviation, on the outcome of COVID-19 inpatients within 15 days.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive inpatient (PCR or other certified test mandatory)
* Inpatient showing at least one of the following criterion: Abnormal respiratory auscultation AND SpO2 < 94% without oxygen therapy, OR Acute Respiratory failure requiring either oxygen therapy or high-flow oxygen therapy or non-invasive respirator and/or invasive respirator.

Exclusion Criteria:

* Inpatient requiring legal protection
* Pregnant or breastfeeding woman
* Intensive care inpatient or patient undergoing surgery

Secondary non inclusion criteria :

- Unintentional blinding removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of clinically improved inpatients between D0 and D14 | 14 day after intervention
  Inpatients are considered as clinically improved if they have gained at least 2 points on the following clinical evaluation scale, or if they went back home
  Clinical evaluation scale :1. Outpatient back to normal activities / 2. Outpatient without normal activities / 3. Inpatient without oxygen therapy / 4. Inpatient with oxygen therapy/ 5. Inpatient requiring either nasal high-flow oxygen therapy or non-invasive respirator or both / 6. Inpatient, requiring either ExtraCorporeal Membrane Oxygenation (ECMO) or invasive artificial respirator, or both / 7. Deceased.

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Marie RANGON, Principal Investigator — Fondation Adolphe de Rothschild
Locations (2):
- France (2):
  - Centre Hospitalier Simone Veil, Beauvais
  - Fondation Adolphe de Rothschild, Paris

REFERENCES:
- [Derived] Rangon CM, Barruet R, Mazouni A, Le Cossec C, Thevenin S, Guillaume J, Leguillier T, Huysman F, Luis D. Auricular Neuromodulation for Mass Vagus Nerve Stimulation: Insights From SOS COVID-19 a Multicentric, Randomized, Controlled, Double-Blind French Pilot Study. Front Physiol. 2021 Aug 2;12:704599. doi: 10.3389/fphys.2021.704599. eCollection 2021. PMID 34408665